CLINICAL TRIAL: NCT04635280
Title: Evaluation of Satisfaction Regarding Home Healthcare Provider (HHP) Management of Type 1 Diabetic Patients Equipped With the "Closed-loop" Automated Insulin Delivery System (or "Artificial Pancreas"), Under Normal Conditions of Use
Brief Title: Evaluation of Satisfaction Regarding Home Healthcare Provider (HHP) Management of Type 1 Diabetic Patients Using a Closed-loop Automatic Insulin Delivery System
Acronym: SATURN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ALMED-19-001
Record Dates: First submitted 2020-11-04; First posted 2020-11-19 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Diabetes type1
Keywords: Artificial pancreas; Patient management; Technical telemonitoring; Home Healthcare Provider
MeSH Terms: interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed-loop automatic insulin delivery system (Experimental): Adults type 1 diabetic patients equipped with a closed-loop automatic insulin delivery system (or artificial pancreas)
  Interventions: Device: any closed-loop automatic insulin delivery system (or artificial pancreas) European Conformity (CE)-marking

INTERVENTIONS:
Device: any closed-loop automatic insulin delivery system (or artificial pancreas) European Conformity (CE)-marking — A closed-loop automatic insulin delivery system includes a combination of an insulin pump, a continuous glucose monitoring system and an algorithm.

SUMMARY:
SATURN study aims at evaluating Home Healthcare Provider (HHP) Management of type 1 diabetic patients using a closed-loop automatic insulin delivery system (or artificial pancreas), and specifically satisfaction and interactions of all people involved (patients, HHPs, hospital healthcare teams) after 1 and 3 months of follow-up, under normal conditions of use.

DETAILED DESCRIPTION:
National, multi-centre, longitudinal, non-comparative interventional study with minimal risks and constraints.

Two French hospitals and their HHP representatives will participate in the study. A recruitment of a total of 35 patients is expected.

Adult type 1 diabetic patients for whom the investigator prescribes the use of a closed-loop automatic insulin delivery system (or artificial pancreas) consisting in an insulin pump with a continuous glucose monitoring system combined with a dedicated terminal.

Patients will be monitored for a period of 3 months, starting from the end of the device installation procedure.

HHP Management comprises three distinct phases: pre-installation, installation and follow-up during which number, nature and duration of contacts (visits/telephone calls) may vary according to patient's needs, investigator's judgement and practice, and judgement of HHP staff.

Pre-installation and installation phases consist of two patients' visits at hospital, and of two to five visits from HHP staff to patients' home (only one visit at hospital). Follow-up phase held after installation consists of four patients' contacts (phone contact and/or home visit) performed by HHP staff.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic patient diagnosed for at least 2 years
* Patient treated with an external insulin pump for at least 6 months
* Patient with an HbA1c level less than or equal to 10% in the past 4 months
* Patient with U100 short-acting insulin (Novorapid or Humalog) requirements between the lower and upper bounds set by the pump of the closed-loop automatic insulin delivery system (or artificial pancreas)
* Patient who is not isolated, who does not live alone or who has a "resource" person living nearby with her/his own telephone and a key to the patient's home
* Patient living in an area covered by a Global System for Mobile Communications (GSM) network and not planning to travel outside France or outside an area covered by a GSM network within 30 days of the closed-loop automatic insulin delivery system (or artificial pancreas) being installed
* Patient at least 18 years old and whose age complies with the eligibility criteria for each medical device of the closed-loop automatic insulin delivery system (or artificial pancreas)
* Patient registered with a Social Security scheme
* Patient who has agreed to comply with the requirements of the study and has signed the free and informed consent form
* Patient who the investigator deems capable of using a closed-loop automatic insulin delivery system (or artificial pancreas) under normal conditions of use.

Exclusion Criteria:

* Patient with any serious pathology that could affect his/her participation in the study
* Patient undergoing treatment that could affect the physiology of diabetes, i.e., that leads to interactions with glucose and/or insulin, in the investigator's judgement
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman
* Absence of contraception deemed effective by the investigator for a woman of child-bearing age
* Psychological and/or physical state which could affect the proper follow-up of the study procedures
* Severe hypoglycaemia which has led to convulsions or a loss of consciousness in the last 12 months
* Decrease in the perceived sensation of hypoglycaemia, in the investigator's judgement
* Altered renal function (creatinine clearance < 30 ml/min measured in the last 6 months)
* Patient who has had a pancreas or pancreatic islet transplant
* Patient with serious uncorrected hearing and/or visual problems
* Patient included in another clinical study or who has taken part in another clinical study in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène HANAIRE, MD, PhD, Principal Investigator — Hôpital de Rangueil - 31059 Toulouse - France
Locations (2):
- France (2):
  - CHU de Nantes - Hôpital Nord Laennec, Nantes
  - CHU de Toulouse - Hôpital Rangueil, Toulouse

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 patients were enrolled from 2 french centres. First Patient Enrolled: 10 May 2021 Last patient Enrolled: 22 September 2021 Last Patient Completed: 12 January 2022
Groups:
- Hybrid Closed-loop Automatic Insulin Delivery System: A closed-loop automatic insulin delivery system includes a combination of an insulin pump, a continuous glucose monitoring system and an algorithm.
Period: Overall Study
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 35
HbA1c in category [Count of Participants; unit: Participants]
  <7% | 10
  7%-<8% | 18
  8%-10% | 7
HbA1c [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 7.35 (0.77)
Time since type 1 diabetes diagnosis [Mean (Standard Deviation); unit: years] — Time between the date of type 1 diabetes diagnosis and the date of inclusion visit, converted in years
  years | 23.3 (12.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Satisfaction Regarding the Management in General, at Day 30 and Day 90, by the CSQ-8 Questionnaire
Description: Satisfaction regarding the management in general was assessed using the Client Satisfaction Questionnaire (CSQ-8). CSQ-8 is a validated questionnaire that measures patients' overall satisfaction with their management in general. It contains 8 questions and each question is answered using a 4-point scale. The score ranges from 8 to 32, with higher values indicating higher satisfaction.
  Patients were considered as satisfied if they reached a score above 20 points.
Time Frame: Day 30 and Day 90
Population: Intention-To-Treat (ITT) population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
Participants
  Patients satisfied - Day 30 | 35
  Patients satisfied - Day 90 | 35

2. Primary Outcome: Number of Participants With Maintenance of Global Patient Satisfaction Regarding the Management in General, at Day 90, by the CSQ-8 Questionnaire
Description: Satisfaction regarding the management in general was assessed using the Client Satisfaction Questionnaire (CSQ-8). CSQ-8 is a validated questionnaire that measures patients' overall satisfaction with their management in general. It contains 8 questions and each question is answered using a 4-point scale. The score ranges from 8 to 32, with higher values indicating higher satisfaction. Satisfaction was defined by a score above 20 points. Maintenance of satisfaction is measured on D90 by a score above 20 points which has not decreased by more than 4 points compared with D30.
Time Frame: Day 90
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
Participants
  Satisfaction maintained | 33
  Satisfaction not maintained | 2

3. Primary Outcome: Description of Patient Satisfaction and Experience Regarding the Management by HHP at Day 30 and Day 90
Description: The questionnaire was developed for the study by the French Diabetes Federation, aiming at evaluating patient satisfaction and experience with their management by the HHP. 16 questions assessed the proactiveness, availability and HHP nurse advice. A global score ranging from 13 to 57 was calculated, with higher values indicating higher satisfaction. The global score was only calculated when all questions were answered.
Time Frame: Day 30 and Day 90
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria All participants completed at least partially the questionnaire; 27 participants completed entirely the questionnaire at D30 and 30 participants completed entirely the questionnaire at D90; 31 participants completed entirely the questionnaire at either D30 or D90.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 31
units on a scale
  Day 30: number analyzed (Participants) | 27
  Day 30 | 47.6 (5.2)
  Day 90: number analyzed (Participants) | 30
  Day 90 | 46.8 (5.3)

4. Secondary Outcome: Total Number of HHP Interactions
Description: Cumulative number of HHP interactions during the study, in total and by type of contact. Unplanned additional contacts are included.
Time Frame: Throughout the study, up to 3 months
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Mean (Standard Deviation); unit: number of contacts
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
number of contacts
  Total number of contacts | 7.3 (1.5)
  Phone contacts | 2.8 (1.5)
  Physical visits contacts | 3.8 (1.1)

5. Secondary Outcome: Cumulative Duration of HHP Interactions
Description: Cumulative duration of HHP interactions during the study, for all contacts and by type of contact
Time Frame: Throughout the study, up to 3 months
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
minutes
  All contacts | 472 (123)
  Phone contacts | 66 (47)
  Physical visits contacts | 329 (97)

6. Secondary Outcome: Comparison of the HHP Observed Management With the Theoretical Management Described in the Medical Device's Information Record.
Description: Number and percentage of patients who required increased follow-up/support, identical follow-up/support and reduced follow-up/ support in relation to what was recommended in the supplier's information record. The maximal number of contacts expected in the supplier's information record was 9 contacts.
Time Frame: Throughout the study, up to 3 months
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
Participants
  Reduced (< 9 contacts) | 29
  Identical (=9 contacts) | 4
  Increased (>9 contacts) | 2

7. Secondary Outcome: Quality of Life Questionnaire (EQ-5D) Summary Index at Inclusion, Day 30 and Day 90
Description: The patient's quality of life was assessed by the quality of life questionnaire (EQ-5D-5L), validated in French Language. It is composed of 5 items each corresponding to a specific dimension (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and divided into 5 levels of perception (1. no problem, 2. slight problems, 3. moderate problems, 4. severe problems, 5. extreme problems/incapacity). The digits for the 5 dimensions were combined in a 5-digit code describing the patient's health state and were converted into a summary index value using the french value sets. The summary index ranges between 0 (dead) and 1 (perfect health)
Time Frame: At inclusion, Day 30 and Day 90
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
units on a scale
  Inclusion | 0.95 (0.10)
  Day 30 | 0.94 (0.09)
  Day 90: number analyzed (Participants) | 34
  Day 90 | 0.94 (0.10)

8. Secondary Outcome: Hypoglycaemia Fear Survey (HFS) Total Score at Inclusion, Day 30 and Day 90
Description: The HFS-II is a validated questionnaire that will be used to measure quality of life and daily constraints with respect to hypoglycaemia-related behaviours and concerns in adults with type 1 diabetes. The HFS total score ranges from 0 to 132, with higher values indicating a higher fear of hypoglycemia.
Time Frame: At inclusion, Day 30 and Day 90.
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
score on a scale
  Inclusion | 31.2 (15.7)
  Day 30 | 25.7 (20.1)
  Day 90 | 23.1 (16.8)

9. Secondary Outcome: Number of Daily Constraints Encountered by Patients on the Past Month at Inclusion, Day 30 and Day 90
Description: The patient's everyday constraints were assessed based on the past month, with a questionnaire in the form of a pre-established multiple-choice list. The questionnaire was developed by the French Diabetes Federation and includes 12 items: - Managing other people's perceptions of my diabetes - Anticipating my activities - Thinking about my diabetes all the time - Dealing with my diabetes all the time - Fear of experiencing hypoglycaemia - Fear of experiencing hyperglycaemia - Uncertainties about my future health - Carrying one or more treatment devices on me at all times - Handling my continuous glucose sensor - Handling all my treatment equipment (pump, glucose sensor, etc.) - Determining my insulin doses several times a day - Hearing the audible alarms of my treatment equipment (pump, glucose sensor, etc.). The number of constraints is reported.
Time Frame: At inclusion, Day 30 and Day 90
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Mean (Standard Deviation); unit: number of constraints ticked
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
number of constraints ticked
  Inclusion | 3.4 (1.8)
  Day 30 | 2.5 (1.2)
  Day 90: number analyzed (Participants) | 34
  Day 90 | 2.9 (1.8)

10. Secondary Outcome: Number of Participants Who Expected and Perceived Benefits With Respect to the Closed-loop Automated Insulin Delivery System at Inclusion and Day 90
Description: The expected and perceived benefits with respect to the closed-loop automated insulin delivery system was assessed by the questionnaire "You and the Hybrid Closed-Loop (HCL) automated insulin delivery system" developed by the French Diabetes Federation for the study.
  Only 2 benefits are presented
Time Frame: At inclusion and Day 90
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
Participants
  Expected experiencing less hypo/ hyperglycemia at Inclusion | 35
  Noticed less hypo/ hyperglycemia at D90 | 31
  Expected spending more time in glycemic target at inclusion | 34
  Noticed spending more time in glycemic target at D90: number analyzed (Participants) | 34
  Noticed spending more time in glycemic target at D90 | 32

11. Secondary Outcome: Beliefs About Medicines Questionnaire (BMQ) Scores at Inclusion and D90
Description: The patient's beliefs about the medical treatment were assessed by the specific section of the BMQ (Beliefs about Medicines Questionnaire), validated in French for diabetes. The specific BMQ consists of two parts: Part one contains five questions related to the need for the treatment and part two contains five questions on concerns about the prescription. The 10 questions are answered using a 5-point scale (1. strongly disagree, 2. disagree, 3. uncertain, 4. agree and 5. strongly agree). The results take the form of two scores ranging from 5 to 25, with higher value indicating higher need/concerns for treatment.
Time Frame: At inclusion and Day 90
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
units on a scale
  BMQ - higher need score at Inclusion | 19.5 (2.3)
  BMQ - higher need score at D90 | 19.1 (2.1)
  BMQ - concerns score at Inclusion | 15.9 (2.3)
  BMQ - concerns score at D90 | 15.8 (2.3)

12. Secondary Outcome: HbA1c at Inclusion and Day 90
Description: HbA1c (%) at inclusion and Day 90
Time Frame: Inclusion and Day 90
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
percentage of glycated hemoglobin
  Hba1c at Inclusion | 7.35 (0.77)
  Hba1c at Day 90 | 6.68 (0.63)
  Absolute change of HbA1c at D90 from inclusion | -0.67 (0.42)

13. Secondary Outcome: Glycemic Variability at Inclusion and Day 90
Description: Glycemic variability assessed by the coefficient of variation (CV)
Time Frame: At inclusion and Day 90
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variation
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
percentage of coefficient of variation
  Glycemic CV at Inclusion: number analyzed (Participants) | 27
  Glycemic CV at Inclusion | 38.7 (5.8)
  Glycemic CV at Day D90 | 34.1 (5.0)
  Absolute change of Glycemic CV at D90 from installation | -4.2 (4.5)

14. Secondary Outcome: Percentage of Time Spent Over a 4-week Period in Glycemic Target Range at Inclusion and Day 90
Description: Percentage of time spent over a 4-week period in glycemic target range, in hypoglycaemia and in hyperglycaemia. Glycemic target range: 70-180 mg/dl, hypoglycaemia: < 70 mg/dl and hyperglycaemia :> 180 mg/dl
Time Frame: At inclusion and Day 90
Population: ITT population: all included patients fitted with the device who met all of the inclusion and exclusion criteria
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
Number analyzed (Participants) | 35
percentage of time
  Time in range 70-180 mg/dl at inclusion | 57.0 (13.3)
  Time in range 70-180 mg/dl at D90 | 71.4 (9.4)
  Time in hypoglycaemia < 70 mg/dl at inclusion | 4.7 (4.6)
  Time in hypoglycaemia < 70 mg/dl at D90 | 2.1 (1.7)
  Time in hyperglycaemia > 180 mg/dl at inclusion | 37.8 (14.9)
  Time in hyperglycaemia > 180 mg/dl at D90 | 26.4 (9.5)

ADVERSE EVENTS:
Time Frame: From the time signed informed consent is obtained until the end of the study for the patient, up to 3 months
Arm/Group | Hybrid Closed-loop Automatic Insulin Delivery System
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 12/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hybrid Closed-loop Automatic Insulin Delivery System (N=35)
Asthenia (General disorders) | 2 (2)
Catheter site erythema (General disorders) | 2 (2)
Catheter site inflammation (General disorders) | 2 (2)
Diabetic ketosis (Metabolism and nutrition disorders) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Ketosis (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the Sponsor can review results communications prior to public release. According to Article R. 5121-13 of the French Public Health Code, the results of the Research may not be published or the subject of written or oral communications by the PI without prior written consent of the Sponsor.The disclosure restriction applies to the Parties during the entire duration of the agreement and as long as the confidential data are not in the public domain.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT04635280/Prot_SAP_000.pdf